CLINICAL TRIAL: NCT02595632
Title: Exhaled Breath Analysis by Secondary Electrospray Ionization (SESI-MS) in Healthy Controls
Brief Title: Breath Analysis in Healthy Controls
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2015-0187
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Exhaled Breath; Mass Spectrometry; Healthy Subjects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy: Healthy subjects with no apparent lung disease and normal lung function testing.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The purpose of this study is to detect a specific profile of breath in healthy subjects by an untargeted metabolomic study using exhaled breath analysis by mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

1. Normal spirometry (forced expiratory volume in 1 second (FEV1) > 80%, forced vital capacity (FVC) > 80%, FEV1/FVC > 70%.).
2. Age between 18 and 90 years at study entry.

Exclusion Criteria:

1. Presence of an active malignancy.
2. Presence of any lung disease (e.g. asthma, chronic obstructive pulmonary disease (COPD), sarcoidosis)
3. Acute inflammatory disease (e.g. common cold) within the last 6 weeks.
4. Acute or chronic hepatic disease.
5. Renal failure or renal replacement therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects will be included according to the predefined inclusion and exclusion criteria. They will be recruited from the general population by printed flyers, newspaper advertisements and personal communication.
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the mass spectrometric exhaled breath pattern of healthy subjects. | 1 day, single measurement, no follow up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland